CLINICAL TRIAL: NCT06331897
Title: Assessment of Bronchial Asthma & Its Exacerbation : the Utility of Laboratory Investigation , Chest Imaging , Pulmonary Function Tests
Brief Title: Bronchial Asthma & Its Exacerbation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ragab Kamel Mohamed, Resident of Pediatrics department, Assiut University
Other Study IDs: Bronchial asthma
Record Dates: First submitted 2024-03-16; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our goals is to assess :

1¬_ the role of spirometer in case of asthma exacerbation 2_hematological parameters (N/L ratio & platelet indices &CRP )in asthma exacerbation for diagnosing and classifying asthma severity and its exacerbation

DETAILED DESCRIPTION:
Bronchial asthma is a chronic inflammatory disease characterized by bronchial hyper-reactivity, reversible airway obstruction, and excessive mucus production that arises from an inappropriate stimulation of the immune system, especially by environmental aeroallergens .Bronchial asthma exacerbations are episodes described by progressive increase in symptoms of cough, wheezing, shortness of breath, and/or chest tightness, with a progressive decrease in lung function . Few tests are being used for diagnosis of asthma, but at present, no established biomarker is available that may be used for diagnosis and prognosis of asthma . Platelet indices and C-reactive protein (CRP) are markers that reflect a systemic inflammatory response . Bronchial obstruction, variable over time and reversible after using bronchodilator is the hallmark of the respiratory function in bronchial asthma. There are patients with "atypical" functional tests or in whom routine tests (spirometry, peak-flowmetry) are not sufficient for asthma diagnosis (thus necessitating more complex functional tests). Pulmonary function evaluation confirms the diagnostic, establishes disease severity and contributes to disease monitoring. Quality criteria verification (e.g. acceptability of the measurements and reproducibility of the parameters) should precede any interpretation . Neutrophilic, eosinophilic, paucigranulocytic or mixed granulocytic types are four various endotypes of asthma [6] depending on cell counts of peripheral blood .

Neutrophilic inflammations have been studied to be associated with a poor asthma control . In addition to persistent asthma symptoms and atopy, they have been reported to be associated with the presence of eosinophilic inflammation in asthmatic patients . Accordingly, NLR increase in asthmatics was considered. However, data related to NLR in Asthmatic patients is inadequate . Though association between asthma and NLR, was discovered by earlier researches in adults, recent researches did not study NLR relation to neutrophilic asthma . So, we aimed to assess the relation of NLR and bronchial asthma severity and to determine NLR discriminative performance between controlled and uncontrolled asthma . Platelet indices, which include the mean platelet volume (MPV), platelet distribution width (PDW), plateletcrit (PCT), and platelet large cell correlated with white blood cells, PaO2, and symptoms duration, and negatively correlated with forced expiratory volume in the first second, symptoms duration, and hs-CRP (P<0.001).

Higher autophagy of neutrophils has been described in many pulmonary disorders as well as neutrophil extracellular traps and exosomes that has been newly studied as deriving from neutrophil . So neutrophils role in pulmonary diseases have been established. Despite pulmonary diseases pathogeneses are being studied widely, there is still more and more to get clarification of the discrepancy and complexity, particularly the contribution of different immune mechanisms in the progress of pulmonary disorders .

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Bronchial asthma Disease
* must be able to applied to spirometer

Exclusion Criteria: patients have 1-other chest diseases 2- diabetes mellitus and hypertension 3- malignancies and hematological disorder 4- valvular lesions , coronaries disease and heart failure 5- autoimmune diseases .

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children group aged (2-18 years old ) who have bronchial asthma and its exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Broncial asthma & its exacerbation : the utility of laboratory investigation , chest imaging , pulmonary function tests | baseline
  to assess : the role of spirometer in case of asthma exacerbation